CLINICAL TRIAL: NCT05953883
Title: Proteogenomic Signatures Analysis In Ovarian Cancer, Longitudinal Modification On Tumor Tissue Before And After Platinum-Based Neoadjuvant Chemotherapy
Brief Title: Proteogenomic Signatures Analysis In Ovarian Cancer
Acronym: PROGENITOR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5288
Record Dates: First submitted 2023-06-21; First posted 2023-07-20 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Tumor Burden; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Participants are prospectively assigned to an intervention consisting of a tumor biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Participants are prospectively assigned to an intervention consisting of a tumor biopsy.
  Interventions: Procedure: Tumor and blood sample

INTERVENTIONS:
Procedure: Tumor and blood sample — Analyzing proteogenomic profiles in order to find individual platinum-induced modifications on tumor tissue of HGSOC according to chemotherapy response score (CRS). Whole genome sequencing (WGS), transcriptomic (RNAseq) and proteomics analyses on OC tissue samples before and after a standard platinum-based chemotherapy will be carried out and correlated to clinical variables.

SUMMARY:
Proteogenomic analysis to detect individual platinum-induced modifications on tumor tissue of HGSC according to chemotherapy response score (CRS), using a combined approach of High resolution liquid chromatography mass Spectrometry based platform (HR-LC-MS/MS and advanced immunometric methods on illumine platform); multiple supervised machine learning algorithms will be used to discover proteogenomic signatures and biological processes associated with platinum modification during the neoadjuvant chemotherapy treatment. These results contribute to precision medicine by building an accurate proteogenomic profile of ovarian cancer, in order to better understand the underlying mechanisms of different chemotherapy response among affected patients.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed advanced International Federation of Gynecology and Obstetrics (FIGO) stage III A or greater epithelial ovarian cancer addressed to neoadjuvant chemotherapy (NACT) and interval debulking surgery (IDS);

Availability of freshly frozen tissue and FFPE tissue from both exploratory laparoscopy (baseline) and IDS;

Age between 18 and 80 years;

Estimated life expectancy of at least 4 weeks;

Signed informed consent

Exclusion Criteria:

Non-serous histology at frozen section;

Patients with a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (> 10 mg equivalent prednisone/daily) or any other form of immunosuppressive therapy within 7 days prior to the enrollment;

Previous diagnosis of cancer within 5 years.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2025-03-17 (Estimated)

PRIMARY OUTCOMES:
DATA CORRELATION | 12 months
  To correlate longitudinal protegenomic data to chemotherapy response score (CRS)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Nero, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy